CLINICAL TRIAL: NCT00979251
Title: A Randomized Open Label Study Comparing the Efficacy, Safety, and Tolerability of Oral Administration of Amantadine and Ribavirin With Oseltamivir Versus Oseltamivir to Influenza A Virus Infected Immunocompromised Subjects
Brief Title: Oral Triple Combination Antiviral Drug Therapy for Treatment of Influenza A in Immunocompromised Subjects
Acronym: PO206
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADS-TCAD-PO206
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Influenza
Keywords: Influenza; Immunocompromised; HIV; History of transplant
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; Amantadine; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADS-8902 (Experimental): Amantadine and Ribavirin administered with Oseltamivir phosphate
  Interventions: Drug: ADS-8902
- Comparator (Active Comparator): Oseltamivir Phosphate
  Interventions: Drug: Oseltamivir Phosphate

INTERVENTIONS:
Drug: Oseltamivir Phosphate — Oseltamivir Phosphate, q8h
  Other Names: Tamiflu
  Arms: Comparator
Drug: ADS-8902 — Amantadine Hydrochloride, Ribavirin administered with Oseltamivir Phosphate, q8h
  Other Names: Amantadine Hydrochloride; Rebetol®; Tamiflu®
  Arms: ADS-8902

SUMMARY:
This Phase 2, open label, randomized study will investigate the virologic benefit, clinical efficacy, safety, and tolerability of amantadine and ribavirin with oseltamivir (TCAD) versus oseltamivir monotherapy for the treatment of all strains of influenza A in immunocompromised adult and pediatric subjects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed influenza A by rapid antigen testing
* Immunocompromised as defined by recent solid organ or hematopoietic transplant, chronic graft vs. host disease, taking at least 2 immunosuppressants, undergoing chemotherapy, taking high dose chemotherapeutics, HIV positive
* Clinical diagnosis of influenza
* Onset of illness within 5 days
* Male and female subjects agree to contraception through 24 weeks after last dose

Exclusion Criteria:

* Received more than 1 dose of antiviral agents
* Critically ill
* Creatinine clearance less than 80 mg/mL
* Females who are pregnant and males whose female partners are pregnant
* Received live attenuated virus vaccine within 3 weeks

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Time to clearing of viral shedding | Baseline, Days 2, 4, 6, 8, 10, 15 and 20

SECONDARY OUTCOMES:
Time to alleviation of influenza clinical symptoms | Baseline, Days 2, 4, 6, 8, 10, 15, 20, 38
Proportion of subjects who enter the study with mild to moderate influenza and progress to severe influenza | Baseline, Days 2, 4, 6, 8, 10, 15, 20, 38
Proportion of subjects with a treatment-sensitive influenza A strain at baseline who develop a resistant strain during treatment | Baseline, Days 2, 4, 6, 8, 10, 15, 20
Safety and tolerability (adverse events (AEs), AEs resulting in treatment discontinuation, and Serious AEs) | Through day 210

CONTACTS AND LOCATIONS:
Locations (23):
- United States (14):
  - Adamas Investigational Site, San Francisco, California
  - Adamas Investigational Site, Hollywood, Florida
  - Adamas Investigational Site, Miramar, Florida
  - Adamas Investigational Site, Pinellas Park, Florida
  - Adamas Investigational Site, Honolulu, Hawaii
  - Adamas Investigational Site, Owensboro, Kentucky
  - Adamas Investigational Site, New Orleans, Louisiana
  - Adamas Investigational Site, Las Vegas, Nevada
  - Adamas Investigational Site, New York, New York
  - Adamas Investigational Site, Rapid City, South Dakota
  - Adamas Investigational Site, Memphis, Tennessee
  - Adamas Investigational Site, Amarillo, Texas
  - Adamas Investigational Site, Seattle, Washington
  - Adamas Investigational Site, Tacoma, Washington
- Australia (5):
  - Adamas Investigational Site, Darlinghurst, New South Wales
  - Adamas Investigational Site, Herston, New South Wales
  - Adamas Investigational Site, Sydney, New South Wales
  - Adamas Investigative Site, Parkville, Victoria
  - Adamas Investigational Site, Melbourne
- Canada (2):
  - Adamas Investigational Site, Edmonton, Alberta
  - Adamas Investigational Site, Toronto, Ontario
- Adamas Investigational Site, Leiden, Netherlands
- Adamas Investigational Site, Singapore, Singapore